





**Study Director UKT** 

Dr. Benjamin Steinhilber University Hospital Tübingen

☐ Benjamin.Steinhilber@med.uni-tuebingen.de

**\*** +49 07071-29-86805

Institute of Occupational and Social Medicine and Health Services Research Wilhelmstraße 27 72074 Tübingen, Germany Medical Director: Prof. Dr. M.A. Rieger

## **Informed Consent Form**

Experimental laboratory study **ADVANCE** – Work Physiological-Biomechanical Analysis of a Passive Exoskeleton to Support Occupational Lifting and Flexing Processes"

Ethical approval number: 617/2018BO2 NCT number at ClinicalTrials.gov: NCT03725982

Date of original document creation: 6 August 2018

The consent to participate in the study is only effective if it is personally signed by a person capable of consent and if it can be revoked informally at any time. The approval is only legally relevant if the study participant has been sufficiently informed.







## Informed Consent Form for study participation to:

Experimental laboratory study **ADVANCE** – Work Physiological-Biomechanical Analysis of a Passive Exoskeleton to Support Occupational Lifting and Flexing Processes

Dr. Benjamin Steinhilber
University Hospital Tübingen
Institute of Occupational and Social Medicine and Health Services Research
Wilhelmstraße 27
72074 Tübingen, Germany

## **Informed Consent Form to Participation of the ADVANCE Study:**

- I confirm that I have been informed about the nature, meaning and scope of the study, in
  particular its objectives and the duration, the course, the benefits as well as the risks and
  side effects of participating in the study,
- I confirm that all questions have been answered to my satisfaction,
- I confirm that I have been informed that participation in the study is completely voluntary and that consent can be withdrawn at any time without reason and without disadvantages,
- I confirm that I can contact the person responsible for the study at any time with questions
  or problems using the contact details given above,
- I confirm that I have been informed, if necessary, about taking out volunteer insurance and about the obligations towards the insurance company,
- I confirm that I have received a copy of the information text and the declaration of consent.

| Study Participant: | | |
|---|---|---|
| Tübingen, date: | Signature | Name of the Participant in block letters |
| Study leader: | | |
| Tübingen, date: | Signature | Name of the Study Leader in block letters (employee of the Institute of Occupational and |





